CLINICAL TRIAL: NCT04850768
Title: Evaluation of (NOD)-Like Receptors CARD Domain-containing 4 Levels in Individuals With Healthy and Periodontal Disease
Brief Title: (NOD)-Like Receptors CARD Domain-Containing 4 Levels in Individuals With Periodontitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Ayse Toraman, Dr, Saglik Bilimleri Universitesi
Other Study IDs: 21-29
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Periodontitis; Gingivitis; Healthy
Keywords: NLRC4
MeSH Terms: conditions — Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva and gingival crevicular fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Periodontitis: Individuals with Periodontitis
  Interventions: Other: Saliva; Other: gingival crevicular fluid
- Gingivitis: Individuals with Gingival Inflammation
  Interventions: Other: Saliva; Other: gingival crevicular fluid
- Healthy: Individuals with Periodontally Healthy
  Interventions: Other: Saliva; Other: gingival crevicular fluid

INTERVENTIONS:
Other: Saliva — individuals' saliva samples will be collected and transferred to eppendorf tubes.
  Until biochemical analysis is carried out will be stored in -80ºC.
  Other Names: sampling
Other: gingival crevicular fluid — GCF samples of individuals will be collected by paper strips and transferred to eppendorf tubes.Until biochemical analysis is carried out will be stored in -80ºC.
  Other Names: sampling

SUMMARY:
NLRC4, an inflammasome , is a cytosolic multiprotein complex involved in the initiation and modulation of the immune response. Periodontitis is a chronic inflammatory disease that can start with localized inflammatory reactions created by the supporting tissues surrounding the teeth against microorganisms and then result in loss of teeth. It has been said that proinflammatory cytokines released in the microenvironment of periodontitis can increase the expression of NLRC4 inflammasome genes. The authors think that NLRC4 may play a role in the periodontitis. The aim of this study is to compare the NLRC4, IL-1β and IL-10 levels of healthy and periodontitis individuals.

DETAILED DESCRIPTION:
Periodontitis is a destructive chronic inflammatory disease that can start with localized inflammatory reactions created by the supporting tissues surrounding the teeth against microorganisms and then result in loss of teeth. Inflammasomes are cytosolic multiprotein complex involved in the initiation and modulation of the immune response.

Interleukine -1β ( IL-1β ) levels are associated with periodontal destruction in the pathogenesis of periodontal disease. Interleukine-10 (IL-10) has been reported to decrease periodontal disease progression rate.

Gingival crevicular fluid shows the cellular response in the periodontium. The most important host-related ingredients are inflammatory markers, including cytokines, enzymes, and interleukins. Saliva analysis is used in the diagnosis of systemic conditions as well as in the diagnosis of oral pathologies.

Both NLRC4 and NLRP3 inflammasomes have been shown to play an important role in the induction of interleukin-1β secretion. Periodontitis is induced by a complex microbial biofilm containing multiple Gram-positive and Gram-negative bacteria (including flagellate microorganisms) capable of activating a large number of NLRs. It has been said that proinflammatory cytokines released in the microenvironment of periodontitis can increase the expression of NLRC4 inflammasome genes. Evidence on the role of inflammasomes in periodontal disease is still very poor. The aim of this study is to compare the NLRC4, IL-1β and IL-10 levels of healthy and periodontitis individuals.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy individuals who does not have a disease under treatment, individuals without regular systemic medication

Exclusion Criteria:

* smoking receiving periodontal treatment in the last 6 months pregnancy menopausal or menstrual period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals will be divided into three different groups, about 20-25 people in each group.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-04-16 (Estimated); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
IL-1β levels | through study completion, an average of 6 months
  saliva and DOS levels
IL-10 levels | through study completion, an average of 6 months
  saliva and DOS levels
NLRC4 | through study completion, an average of 6 months
  saliva and DOS levels

SECONDARY OUTCOMES:
Plaque Index | up to 20 weeks
  Silness-Löe
Probing Depth | up to 20 weeks
  millimeter
Bleeding on Probe | up to 20 weeks
  Ainamo&Bay

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Toraman, Dr, Principal Investigator — Saglik Bilimleri Universitesi; Ebru Sağlam, Dr, Study Chair — Saglik Bilimleri Universitesi; Serhat Köseoğlu, assoc prof, Study Chair — Saglik Bilimleri Universitesi; Mehmet Sağlam, assoc prof, Study Chair — Izmir Katip Celebi University; Levent Savran, PhD, Study Chair — Izmir Katip Celebi University
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No